CLINICAL TRIAL: NCT06275490
Title: Evaluation of Post Extraction Hard Tissue Changes Following Ridge Preservation Using Partially Demineralized Dentin Block Versus L- PRF Block in the Esthetic Zone: A Randomized Controlled Pilot Trial
Brief Title: Post Extraction Changes Following Ridge Preservation Using Partially Demineralized Dentin Block Versus L- PRF Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed Mohammed Alhazmi, Principal Investigator Alaa Ahmed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181123PER6_3_1
Record Dates: First submitted 2024-01-12; First posted 2024-02-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Socket Preservation
Keywords: Socket Preservation; L-PRF block; Xenograft

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Pilot Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially Demineralized Dentin Block (Experimental): The extracted tooth will undergo grinding using the tooth transformer device. The produced dentin graft will be of a particle size 400-800 μm. Afterwards.
  -Prepare the partially demineralized dentin block, the L-PRF membranes will be cut into small pieces and mixed with the dentin particles at a ratio of 2 membranes to 0.5 g of dentin, providing a 1:1 volume ratio. The liquid fibrinogen will be added to the homogeneous mixture, and while shaping the mixture into the desired form it will be gently stirred for approximately 10 seconds. Within a few minutes, the fibrinogen will convert into fibrin primarily from the activated blood platelets in the chopped L-PRF membranes. This process will effectively trap the biomaterial and the L-PRF pieces, forming a sturdy block known as the "dentin block," which serves as a convenient and compact graft .The extracted socket will be filled with partially demineralized autogenous dentin graft.
  Interventions: Biological: Partially Demineralized Dentin Block; Biological: L-PRF block
- L- PRF Block (Active Comparator): The same procedure will be performed for preparing the L-PRF block by mixing the L-PRF membranes with xenograft. In both groups, the placed graft will be covered with a L-PRF membrane .The L-PRF clots obtained after 12 min of centrifugation will be placed in the Xpression box (IntraSpin, Intra-Lock, Florida, USA) for 5 min to gently compress (by gravity) into membranes.
  Finally, tension free wound closure will be attained after periosteal releasing incision and suturing using 5/0 proline interrupted sutures.
  An immediate postoperative CBCT scan will be done following the surgical procedure.
  Interventions: Biological: Partially Demineralized Dentin Block; Biological: L-PRF block

INTERVENTIONS:
Biological: Partially Demineralized Dentin Block — The extracted tooth will undergo grinding using the tooth transformer device. The produced dentin graft will be of a particle size 400-800 μm. Afterwards.
  -Prepare the partially demineralized dentin block, the L-PRF membranes will be cut into small pieces and mixed with the dentin particles at a ratio of 2 membranes to 0.5 g of dentin, providing a 1:1 volume ratio. The liquid fibrinogen will be added to the homogeneous mixture, and while shaping the mixture into the desired form it will be gently stirred for approximately 10 seconds. Within a few minutes, the fibrinogen will convert into fibrin primarily from the activated blood platelets in the chopped L-PRF membranes. This process will effectively trap the biomaterial and the L-PRF pieces, forming a sturdy block known as the "dentin block," which serves as a convenient and compact graft .The extracted socket will be filled with partially demineralized autogenous dentin graft.
Biological: L-PRF block — The same procedure will be performed for preparing the L-PRF block by mixing the L-PRF membranes with xenograft. In both groups, the placed graft will be covered with a L-PRF membrane .The L-PRF clots obtained after 12 min of centrifugation will be placed in the Xpression box (IntraSpin, Intra-Lock, Florida, USA) for 5 min to gently compress (by gravity) into membranes.

SUMMARY:
* The aim is to evaluate post extraction hard tissue changes following ridge preservation using partially demineralized dentin block versus L-PRF block in intact socket in the esthetic zone.
* The main question: In patients with un restorable tooth, Will ridge preservation using partially demineralized dentin block be more effective than L-PRF block in managing the post extraction hard tissue alterations?
* After enrolment, periodontal and radiographic examination and patients with badly un-restorative tooth in the esthetic zone will be identified. These patients will undergo to mesio-distal distance between adjacent teeth, corono-apical height of bone, presence of labial undercut, dehiscence, or fenestration and Relation to adjacent teeth measurements using trans gingival probing technique, and preapical radiograph or CBCT .
* In both groups, the desired tooth will be extracted under local anesthesia using peritomies and surgical forceps.
* In intervention group: the teeth will be cleaned and dried, and then the dentin will be ground to obtain particles of a certain size then partially demineralize dentin will obtained by using a tooth transformer machine. At the same time, blood samples are collected and processed to obtain fibrin membranes rich in platelets and leukocytes. This tissue is then mixed with partially demineralized dentin to create a solid mass called a "dentin block". During the process of preserving the alveolar bumps after extraction, this solid mass "dentin mass" is placed inside the dental pockets and covered with fibrin membranes rich in platelets and white blood cells, then 5/0 proline suture are used to fix the fibrin membranes and dentin mass in place. After the recovery period "4-6 months", a biopsy is taken for some cases from the site of the operation for histological evaluation during implant placement.
* In control group: the same steps as the first group will be used, but by replacing the partially demineralized dental graft with a xenograft.
* Outcomes: Radiographic vertical buccal bone changes, vertical Palatal bone changes, horizontal bone changes, Percentage of new vital bone formation, Percentage of residual bone graft, Implant Primary Stability. The results directly postoperative and 4-6 months postoperatively.

DETAILED DESCRIPTION:
* Objective of the study: aims to evaluate post extraction hard tissue changes following ridge preservation using partially demineralized dentin block versus L-PRF block in intact socket in the esthetic zone.
* Research Procedure:

Patients will be selected from the outpatient clinic of the Oral Medicine and Periodontology Department, Faculty of Dentistry, Cairo University.

- General operative procedures: The patients who fulfil the inclusion criteria will be enrolled. The nature of the study will be explained to each patient as well as the importance of compliance with pre- and post-operative instructions and follow-up visits. Each patient will be asked to sign an informed consent (appendix 1). After enrolment, periodontal and radiographic examination and patients with badly un-restorative tooth in the esthetic zone will be identified. These patients will undergo to mesio-distal distance between adjacent teeth, corono-apical height of bone, presence of labial undercut, dehiscence, or fenestration and Relation to adjacent teeth measurements using trans gingival probing technique, and preapical radiograph or CBCT .

- Initial Therapy: The initial therapy will consist of periodontal treatment (phase I therapy) including supra-gingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques.

* Atraumatic extraction:

  * Local anaesthesia will be administered via buccal and palatal infiltration prior to any surgical procedure.
  * In both groups, flapless atraumatic tooth extraction will be performed which includes an intrasulcular incision using a 15c blade, then a periotome is inserted between the root and the surrounding bone in a wedging action all sides around the root. Afterwards, a small sized straight elevator will be used to luxate the root and a remaining root forceps will be used to deliver it. Lucas curette will be used to clean the extraction socket of any apical pathology and granulation tissue.
* In intervention group, the partially demineralized dentin graft will be prepared as follows:

  ✓ The extracted tooth will be decontaminated and cleaned with a diamond bur under abundant irrigation with physiological water. All filling materials (gutta-percha, composite, luting cements, etc.) will be removed with the outmost care. Subsequently, the tooth will be cut into fragments (5 × 5 mm) and will be dried using air and ground with the Tooth Transformer device following the manufacturer's protocol. Dentin particles will be obtained with a dimension of 400 - 800 μm.
* L-PRF membranes will be prepared as follows:

  * Partially demineralized dentin particles will be obtained with a dimension of 300-1200 μm.

At the same time, L-PRF membranes will be prepared. Four 10-cc blood samples will be collected in vacutainer tubes without anticoagulant (red cap, glass coating) and immediately centrifuged at 2700 rpm (408g) for 12 min (IntraSpin, Intra- Lock, Florida, USA).

* Two extra blood samples will be collected in 9-cc non-coated vacutainer tubes also without anticoagulants (white cap). These last samples will be centrifuged at 2700 rpm for 3 min only. The yellow fluid (liquid fibrinogen) at the top of the white cap tubes will be aspirated with a sterile syringe, avoiding red blood cells.
* The L-PRF clots obtained after 12 min of centrifugation will be placed in the Xpression box (IntraSpin, Intra-Lock, Florida, USA) for 5 min to gently compress (by gravity) into membranes.

To prepare the partially demineralized dentin block, the L-PRF membranes will be cut into small pieces and mixed with the dentin particles at a ratio of 2 membranes to 0.5 g of dentin, providing a 1:1 volume ratio. The liquid fibrinogen will be added to the homogeneous mixture, and while shaping the mixture into the desired form, it will be gently stirred for approximately 10 seconds.

Within a few minutes, the fibrinogen will convert into fibrin primarily from the activated blood platelets in the chopped L-PRF membranes. This process will effectively trap the biomaterial and the 16 L-PRF pieces, forming a sturdy block known as the "dentin block," which serves as a convenient and compact graft.

* Alveolar ridge preservation:

  * After socket debridement, each socket will be carefully filled with "dentin blocks" that are shaped to match the individual size and contours of each socket. Once the grafts are properly adapted to the sockets, they will be covered with two layers of L-PRF membranes extending 2 mm in the envelope prepared between the periosteum and the bony borders of the socket (360° around).
  * The wound will be secured using 5/0 proline interrupted sutures, not with the intention to close the wound, but simply to keep the graft and membranes stable in position.
* In the control group: The same procedure will be performed for preparing the L-PRF block by mixing the L-PRF membranes with xenograft.
* Biopsy collection:

After a 4-months healing period, at the moment of the implant placement, a biopsy from the core of the grafted site will be obtained using a 2-mm trephine bur. The biopsy will be immediately fixed in 10% neutral buffered formalin and then dehydrated through baths of progressively more concentrated (from 50 to 100%) alcohol and subsequently embedded in paraffin. Finally, a tissue section of 4-μm thick will be prepared and stained with hematoxylin-eosin for histological analysis.

- Late implant placement:

* After complete bone healing of the extraction socket 4 -6 months following tooth extraction, late implant placement will be performed.
* Local anesthesia in which Septocaine (Articaine hydrochloride 4% with 1:100000 Epinephrine) will be administered via buccal and palatal infiltration prior to any surgical procedure.
* In some cases, from both groups, a triangular flap design will be used which involves a midcrestal horizontal incision with an intrasulcular incision on each distal tooth to the edentulous area. Then, 2 vertical releasing incision will be made at the line angles of the adjacent teeth. This will be followed by full thickness flap elevation.
* Implant osteotomy will then be prepared using sequential drilling according to the manufacturer instructions, to allow implant placement in proper 3D prosthetic position. Finally, implant will be inserted into the prepared osteotomy.

Outcomes: Radiographic vertical buccal bone changes, vertical Palatal bone changes, horizontal bone changes, Percentage of new vital bone formation, Percentage of residual bone graft, Implant Primary Stability.

The results directly postoperative and 4-6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Healthy individuals with no medical history.
* Patients who have a single non-restorable tooth in the esthetic zone.
* Post-extraction socket with four bone walls, the buccal plate is partially missing following extraction of the tooth. (Type II Extraction socket).
* Patients capable of understanding or signing the informed consent form before surgery and capable of meeting oral cleaning requirements for implant placement.

Exclusion Criteria:

* Systemic disease that might impair bone metabolism, antiresorptive therapy (as bisphosphonates),pregnancy, psychiatric conditions.
* Heavy smokers (> 10 cigarettes)
* The presence of acute or chronic infection at the site of tooth extraction with lack of treatment for periodontal disease, or x-rays showing loss of alveolar bone on the adjacent teeth.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Radiographic vertical bone changes | after 4-6 months of the surgery
  CBCT scans will be performed at baseline and 4-6 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish reference,the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn.

SECONDARY OUTCOMES:
Radiographic horizontal bone changes | after 4-6 months of the surgery
  CBCT scans will be performed at baseline and 4- 6 months postoperatively.
Percentage of new vital bone formation and residual graft | after 4-6 months of the surgery
  The biopsies will be stored in a 10% formalin solution for preservation. Afterward, they will undergo decalcification in EDTA for a duration of four weeks. Following decalcification, the specimens will be processed and embedded in paraffin to create tissue blocks. Longitudinal sections of 5μm thickness will be cut from the paraffin blocks. These sections will be stained using hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains for histological evaluation and histomorphometric analysis. Photomicrographs of the stained sections will be captured using a digital light microscope (Leica Digital Microscope, Leica Microsystems, Germany).
Implant Primary Stability | after 4-6 months of the surgery
  will be assessed using the Osstell Mentor Resonance Frequency Analyzer (Osstell AB, Goteborg, Sweden). Two measurements will be taken in the buccolingual and mesiodistal directions for each implant. The average of these two measurements will be recorded as the representative implant stability quotient (ISQ) for each individual implant.

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University
Locations (1):
- Faculty of dentistry Cairo University, Cairo, Elmanil, Egypt